CLINICAL TRIAL: NCT04718779
Title: A Multicenter, Interventional, Retrospective and Prospective Study of Enzyme Replacement Therapy (VPRIV) Clinical Outcomes and Safety in Gaucher Disease Type 1 Patients Previously Treated With Substrate Reduction Therapy
Brief Title: A Study of Enzyme Replacement Therapy (VPRIV) in People With Type 1 Gaucher Disease Who Were Previously Treated With Substrate Reduction Therapy
Acronym: SWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-669-4017
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Prospective (Experimental): Participants with Gaucher's Disease 1 (GD1) transitioning from SRTs to ERT (VPRIV) or ERT to SRT and then to ERT (VPRIV) in a real-world setting among adults 18 and older will be studied by observing standard patient care and by reviewing the results of tests and assessments that would be performed as part of their routine treatment.
  Interventions: Other: Digital Engagement Application (GD App)
- Arm B: Retrospective (Experimental): Participants with GD1 transitioning from SRT to ERT (VPRIV) or ERT to SRT and then to ERT (VPRIV) previously (within the past 5 years at the time of enrollment) will be assessed retrospectively after switch to ERT for up to 12 months.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: Digital Engagement Application (GD App) — This is a chart review (prospective) data analysis study to describe the effect of the treatment change on the clinical parameters and patient reported outcomes (PROs) with the use of a digital engagement application (GD app) (to evaluate participants clinical engagement, shared decision making, emotional wellbeing, activities of daily living, goal attainment and Gaucher Disease specific measures).
  Arms: Arm A: Prospective
Other: No Intervention — This is a chart review (retrospective) data analysis study to describe the effect of the treatment change on the clinical parameters.
  Arms: Arm B: Retrospective

SUMMARY:
The study will provide information on outcomes in people with type 1 Gaucher disease when they are treated with velaglucarase alfa (also called VPRIV), under standard care. Standard care means the participant will be treated according to the clinic's standard practice. The study sponsor will not be involved in how participants are treated with VPRIV, will provide instructions on how the clinic will record what happens during the study.

VPRIV is a type of enzyme replacement therapy (also known as ERT). Before starting the study, participants must either have switched from substrate reduction therapies (SRT) to VPRIV or switched from other enzyme replacement therapies to SRT then finally to VPRIV. During this time, medical data will be collected from the participants' medical records.

During the study, participants will be treated with VPRIV according to their clinic's standard practice. VPRIV is given by a slow injection into the vein, also known as an infusion. This will happen in the clinic or at home.

The study will record if blood levels of specific substances remain stable or improve during the switch to treatment with VPRIV. Some of these substances will show if organs such as the liver or spleen are working well. Others are blood cells that help blood to clot, known as platelets. Another is a substance in a red blood cell used to carry oxygen around the body, known as hemoglobin.

Participants will use a digital tool so they can be more involved in decision making in their treatment. The digital tool is a mobile phone app, in which each participant can log their daily activities, their general health and wellbeing, and other key information.

Medical data will also be collected from the participants' charts during this time.

Health problems of the participants will be recorded during the study to check if there were any side effects from VPRIV treatment.

Participants will be in this study for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

Participant eligibility is determined according to the following criteria prior to entry into the study:

* In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
* Participant either signs and dates a written, informed consent form or completes an e-consent process prior to the initiation of any study procedures.
* Participant has been diagnosed with GD type I; diagnosis was confirmed biochemically and/or genetically.
* Participant has been treated with SRT for at least 3 months prior to switch to VPRIV.
* Participant has been treated with VPRIV at least 3 months prior to enrollment (Baseline [Day 0]).
* Participant is aged 18 or older.
* Arm A: Participant is able to use mobile application based on clinician's judgment, (e.g., owns an iPhone version 5 or later or smartphones with Android operating systems, have an active data plan or regular Wi-Fi access).
* Arm A: The participant's primary language is English.

Exclusion Criteria:

Any participant who meets any of the following criteria will not qualify for entry into the study:

* Participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
* Participant is judged by the investigator as being ineligible for any other reason.
* Participant has L444P/L444P GBA1 genotype (c.1448T greater than [>] C).
* Participant has Parkinson's disease, a history of central nervous system [CNS] manifestations, or any other neurological disorder (e.g. Lewy Body Disease, Alzheimer's Disease, Amyotrophic Lateral Sclerosis, Multiple sclerosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- The Lysosomal and Rare Disorders Research and Treatment Center, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/600e8a40565ce300294c6ae6

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 sites in United States from 22 April 2021 to 16 February 2023.
Pre-assignment Details: A total of 4 participants were enrolled in the study. This is an interventional, retrospective and prospective study to describe the effect of the treatment change on the clinical parameters and patient reported outcomes (PROs) with the use of a digital engagement application.
Groups:
- Arm A: Prospective: Participants with Gaucher's Disease 1 (GD1) who were treated with substrate reduction therapy (SRT) for at least 3 months before being switched to enzyme replacement therapy (ERT) velaglucerase alfa (VPRIV) were followed-up prospectively for 12 months from the switch from SRT to ERT (baseline). All participants were treated in accordance with physician treatment plan (standard clinical practice).
- Arm B: Retrospective: Participants with GD1 transitioning from SRT to ERT (VPRIV) or ERT to SRT and then to ERT (VPRIV) previously (within the past 5 years at the time of enrollment) were followed-up retrospectively for up to 12 months before being switched from SRT to ERT (VPRIV). All participants were treated in accordance with physician treatment plan (standard clinical practice).
Period: Overall Study
Arm/Group | Arm A: Prospective | Arm B: Retrospective
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose medical charts were retrieved and observed in this study. Only 4 participants were enrolled in this study. Based on the low enrolment number, "Overall Arm" data was collected and reported in order to protect and maintain participant privacy/confidentiality.
Groups:
- All GD1 Participants: All participants with GD1 who were treated with SRT for at least 3 months before being switched to ERT (VPRIV) were followed-up prospectively for 12 months from the switch from SRT to ERT (baseline); and participants transitioning from SRT to ERT (VPRIV) or ERT to SRT and then to ERT (VPRIV) previously (within the past 5 years at the time of enrollment) were followed-up retrospectively for up to 12 months before being switched from SRT to ERT (VPRIV). All participants were treated in accordance with physician treatment plan (standard clinical practice).
Arm/Group | All GD1 Participants
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (22.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Stable Hemoglobin (Hb) Concentration From Baseline up to Month 12
Description: Hemoglobin concentration level was assessed from the blood sample. Clinical stability from baseline was calculated using prespecified threshold of hemoglobin concentration level less than (<) 1.5 gram per deciliter (g/dl) decrease level. Number of participants with clinically stable hemoglobin from baseline up to Month 12 were reported.
Time Frame: From Baseline up to Month 12
Population: Analysis population included all eligible participants whose medical charts were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Prospective: Participants with GD1 who were treated with SRT for at least 3 months before being switched to ERT (VPRIV) were followed-up prospectively for 12 months from the switch from SRT to ERT (baseline). All participants were treated in accordance with physician treatment plan (standard clinical practice).
Arm/Group | Arm A: Prospective | Arm B: Retrospective
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Primary Outcome: Number of Participants With Clinically Stable Platelet Count From Baseline in Platelet Count up to Month 12
Description: Platelet count concentration level was assessed from the blood sample. Clinical stability from baseline was calculated using prespecified threshold of platelet count < 25 percent (%) decrease levels. Number of participants with clinically stable platelet count from baseline up to Month 12 were reported.
Time Frame: From Baseline up to Month 12
Population: Analysis population included all eligible participants whose medical charts were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Prospective | Arm B: Retrospective
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

3. Primary Outcome: Number of Participants With Clinically Stable Liver Volume From Baseline up to Month 12
Description: Clinical stability from baseline was calculated using prespecified threshold of liver volume < 20 % increase, was assessed using ultrasound or Magnetic Resonance Image (MRI). Number of participants with clinically stable liver volume from baseline up to Month 12 were reported.
Time Frame: From Baseline up to Month 12
Population: Data for this outcome measure could not be collected and analyzed as no participants were evaluable for the specified parameter.
Arm/Group | Arm A: Prospective | Arm B: Retrospective
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Stable Spleen Volume From Baseline up to Month 12
Description: Clinical stability from baseline was calculated using prespecified threshold of spleen volume < 25 % increase was assessed using ultrasound or MRI. Number of participants with clinically stable spleen volume from baseline up to Month 12 were reported.
Time Frame: From Baseline up to Month 12
Population: as for outcome 3
Arm/Group | Arm A: Prospective | Arm B: Retrospective
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered with a drug; it does not necessarily have to have a causal relationship with the treatment. An SAE was any event that resulted in: death; was life-threatening; required inpatient hospitalization or resulted in prolongation of existing hospitalization; persistent or significant disability/incapacity; was a congenital anomaly/birth defect or a medically important event. AEs included both SAEs, and non-serious AEs.
Time Frame: From start of the study up to Month 12
Population: Analysis population included all eligible participants whose medical charts were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Prospective | Arm B: Retrospective
Number analyzed (Participants) | 2 | 2
Participants
  Participants with AEs | 0 | 0
  Participants with Serious AEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of the study up to Month 12
Arm/Group | Arm A: Prospective | Arm B: Retrospective
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04718779/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT04718779/SAP_002.pdf